CLINICAL TRIAL: NCT03213548
Title: Aesthetic and Functional Results of Alar Base Modifications in Rhinoplasty : A Randomized Clinical Trial
Brief Title: Aesthetic and Functional Results of Alar Base Modifications in Rhinoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59622316.0.0000.5327
Record Dates: First submitted 2017-06-28; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Rhinoplasty; Surgical Procedure, Unspecified; Surgery, Plastic; Cicatrix; Healing Scar
Keywords: alar base reduction; alar facial groove; alectomy; Flare; Nose
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: double blind clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alar facial groove Incision (Experimental): Alar Base surgical modification with surgical inions in the alar facial groove
  Interventions: Procedure: Alar facial groove incision
- Alar facial groove spared (Active Comparator): Alar Base surgical modification with surgical incisions 1mm above the alar facial groove
  Interventions: Procedure: Alar facial groove spared

INTERVENTIONS:
Procedure: Alar facial groove incision — All procedures related to alterations in the alar base will be based on an algorithm proposed by 2010 Adamnson et al lar Soft-Tissue Techniques in Rhinoplasty Algorithmic Approach, Quantifiable Guidelines, and Scar Outcomes From a Single Surgeon Experience ,published at Archives Facial Plastic Surgery in which a sequential approach is used, evaluating step-by-step surgical needs. Initially, the alar base can be reduced by removing tissue from the nasal sill. At this step, modifications at the shape or the width of the nostrils can be done. After that, a rotation-advancement flap is made, and the sill defect is closed. The nasal flair is then assessed and tissue from the alar border can be removed if needed. The incisions not spare the alar facial groove.
  Arms: Alar facial groove Incision
Procedure: Alar facial groove spared — The technique is the same of the Alar facial groove incision intervention group, but the incisions spare the groove. The incisions will be at 1 mm above the groove.
  Arms: Alar facial groove spared

SUMMARY:
Rhinoplasty is among the most accomplished aesthetic procedures in Plastic Surgery. The mastery of Alar Base modifications is essential for superior aesthetic results. The main indication is to reduce nasal width when it exceeds the intercanthal distance in Caucasian women. Other indications are the modification of the shape of the nostrils or to reduce alar flare in noses with too convex alar base. Since Wier's first description, a series of techniques has been developed with a common goal of making the basal view of the nose close to an equilateral triangle. The location and amount of tissue to be removed will be according to the preoperative or intraoperative indication due to changes in the alar base resulting from reductions in the projection of the nasal tip. One of the controversies in the literature is in the position of the incision in alar base modifications. Some authors prioritize incisions that do not violate the alar facial groove , since the groove region presents a greater number of sebaceous glands, leading to poor scarring results. Other authors have argued that incisions above the sulcus have caused more evident scars, anda that poor healing results would be more associated with aggressive resections of border and bad closing skin techniques.

Due to divergence in the literature, the present study aims to compare, through a double blinded randomized clinical trial, two techniques of alar base modifications that will differentiate only by violating or not the alar facial groove.

DETAILED DESCRIPTION:
The study was performed at the Otorhinolaryngology service Clinicas Hospital of Porto Alegre ( HCPA). Patients who meet the inclusion and exclusion criteria will be invited to participate in the study. All patients who agree to participate in the study, filling out an Informed Consent Form, will have their preoperative consultation registered. Pre- and postoperative follow-up will be performed at the otorhinolaryngology service of HCPA. Patients will be allocated randomly in the intervention and control groups, in blocks of 6, using a computer generated random sequence of numbers. . The allocation will be kept confidential for the patient and for the researchers responsible for measuring the outcomes. intervention group will be submitted to surgical modification of the alar base with incisions in the alar facial groove, the control group will be submitted to a similar technique, but it will save groove.

The surgical technique will be based on a sequential approach based on the 2010 publication Adamnson et al in the Archives of Facial Plastic Surgery "Alar Soft-Tissue Techniques in Rhinoplasty Algorithmic Approach, Quantifiable Measurement of outcomes will be performed by trained and blinded research team members for intervention allocation. Patients will be evaluated at the preoperative visit, and will return to consultations on days 7, 14.30, 60, 90.360 postoperative days, when they will be photographed at the incidences, frontal, ¾ profile, basal, between tip with Eyebrows. At the base line and at 90 postoperative days the following outcomes will be measured: Stony Brook Scale , ROE Scale, Visual Analogue Scale - Satisfaction with aesthetic aspect of the nose, Visual Analogue Scale Intensity of nasal obstruction and NOSE Scale For the comparison of continuous variables will be compared using Student's t test for independent samples or Mann-Whitney non-parametric test, when appropriate. Multivariate analysis will be performed to control confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients from The Department of Otolaryngology of HCPA Hospital who are candidates for functional and / or aesthetic rhinoplasty over 16 years of age, with an indication of alar base modification, will be candidates for the study.

The alar base modification is indicated when the columella-alar distance is greater than the intercanthal distance, when there is presence of asymmetries between the nostrils or its size is too width. In corrections of overprojected noses, there may be enlargement of the base of the alar, with an indication of reduction of the width of the alar at the end of the procedure.

Exclusion Criteria:

* Patients who present (1) Previous alar base surgery modification ; (2) keloid / hypertrophic scar history and (3) Patients with cheek - alar border obtuse angle

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2019-09-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Stony Brook Scar Evaluation Scale (SBSES) | 90 days
  Patients will be evaluated personally by blinded examiners who will graduate the scars according to the standardized Stony Brook scoring evaluation scar which has a minimum score of 0 and a maximum score of 5 points according to 5 characteristics of the scar ( width, height, color, hatch/suture mark, overall appearance)

SECONDARY OUTCOMES:
Rhinoplasty Outcome Evaluation (ROE) Scale | base line and 90 posoperative days
  The Rhinoplasty Outcome Evaluation (ROE) scale is an easy-to-use questionnaire, designed for the evaluation of rhinoplasty results. This instrument is composed of six questions that assess three domains of quality of life: physical, mental / emotional and social. Each question is scored on a scale of 0 to 4 and converted to a total score of 0 to 100, dividing the value by 24 and multiplying by 100. A score above 85 is considered excellent and generally means that the patient is very satisfied. However, the comparison of pre and postoperative values usually provide the most relevant information. Patients will be asked to respond to this scale in the base line and at 90 postoperative days.
Visual Analogue Scale - Satisfaction with aesthetic aspect of the nose | base line and 90 posoperative days
  Patients will be asked to complete an analogue-visual scale (Annex 3) indicating the degree of satisfaction with the appearance of their nose. This scale will be converted into a scale ranging from 0 to 10, and the value 10 represents the highest satisfaction level possible. The scale will be applied in the base line as well as in the 90 postoperative days.
Intensity of nasal obstruction | base line and 90 posoperative days
  Patients will be asked to complete an analogue-visual scale indicating the severity of their nasal obstruction that will be converted from 0 to 10, and the value 10 represents symptoms of nasal obstruction of greater intensity. The scale will be applied at the base line, as well as at the 90 postoperative days.
NOSE Scale | base line and 90 posoperative days
  The NOSE (Nasal Obstruction Symptom Evaluation Scale) scale will be used to measure the quality of life related to nasal obstruction. It is a validated instrument specifically designed for use in patients with nasal obstruction. According to this scale patients are asked to evaluate difficulty breathing in a general way and specifically the difficulty in breathing through the nose, breathing during sleep, and severity of their nasal congestion. The severity of the symptoms is recorded on a scale of 0 to 4, with 0 being the absence of a problem and 4 being a serious problem. The possible scores range from 0 to 20 and the higher scores indicate a higher degree of nasal obstruction. The sum of the scores is multiplied by 5 so as to obtain a final score ranging from 0 to 100, with higher values associated with poorer quality of life.
  The scale will be applied at the base line and at 90 postoperative days.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lavinsky, PHD, Principal Investigator — Porto Alegre Clinicas Hospital ( HCPA)
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rohrich RJ, Ahmad J. Rhinoplasty. Plast Reconstr Surg. 2011 Aug;128(2):49e-73e. doi: 10.1097/PRS.0b013e31821e7191. PMID 21788798
- [Background] Kridel RW, Castellano RD. A simplified approach to alar base reduction: a review of 124 patients over 20 years. Arch Facial Plast Surg. 2005 Mar-Apr;7(2):81-93. doi: 10.1001/archfaci.7.2.81. PMID 15781717
- [Background] Warner JP, Chauhan N, Adamson PA. Alar soft-tissue techniques in rhinoplasty: algorithmic approach, quantifiable guidelines, and scar outcomes from a single surgeon experience. Arch Facial Plast Surg. 2010 May-Jun;12(3):149-58. doi: 10.1001/archfacial.2010.30. PMID 20479430
- [Background] Bennett GH, Lessow A, Song P, Constantinides M. The long-term effects of alar base reduction. Arch Facial Plast Surg. 2005 Mar-Apr;7(2):94-7. doi: 10.1001/archfaci.7.2.94. PMID 15781718
- [Background] Weir RF. On restoring sunken noses without scarring the face. 1892. Aesthetic Plast Surg. 1988 Nov;12(4):203-6. No abstract available. PMID 3068968
- [Background] Patel AD, Kridel RW. African-American rhinoplasty. Facial Plast Surg. 2010 May;26(2):131-41. doi: 10.1055/s-0030-1253499. Epub 2010 May 4. PMID 20446207
- [Background] Foda HM. Nasal base narrowing: the combined alar base excision technique. Arch Facial Plast Surg. 2007 Jan-Feb;9(1):30-4. doi: 10.1001/archfaci.9.1.30. PMID 17224485
- [Background] Boyette JR, Stucker FJ. African American rhinoplasty. Facial Plast Surg Clin North Am. 2014 Aug;22(3):379-93. doi: 10.1016/j.fsc.2014.04.004. PMID 25049123
- [Background] Stucker FJ, Lian T, Sanders K. African American rhinoplasty. Facial Plast Surg Clin North Am. 2005 Feb;13(1):65-72. doi: 10.1016/j.fsc.2004.04.010. PMID 15519928
- [Background] Porter JP. The average African American male face: an anthropometric analysis. Arch Facial Plast Surg. 2004 Mar-Apr;6(2):78-81. doi: 10.1001/archfaci.6.2.78. PMID 15023793
- [Background] Tardy ME Jr, Patt BS, Walter MA. Alar reduction and sculpture: anatomic concepts. Facial Plast Surg. 1993 Oct;9(4):295-305. doi: 10.1055/s-2008-1064623. No abstract available. PMID 8181769
- [Background] Hagan KF. Clinical photography for the plastic surgery practice--the basics. Plast Surg Nurs. 2008 Oct-Dec;28(4):188-92; 193-4. doi: 10.1097/01.PSN.0000342822.44387.c5. PMID 19092585
- [Background] Swamy RS, Sykes JM, Most SP. Principles of photography in rhinoplasty for the digital photographer. Clin Plast Surg. 2010 Apr;37(2):213-21. doi: 10.1016/j.cps.2009.12.003. PMID 20206739
- [Result] Lima LF, Arroyo HH, Jurado JR. Update in alar base reduction in rhinoplasty. Curr Opin Otolaryngol Head Neck Surg. 2016 Aug;24(4):316-21. doi: 10.1097/MOO.0000000000000277. PMID 27261942